CLINICAL TRIAL: NCT06555497
Title: A Pilot Study of Topical 1% Methotrexate Gel Versus Clobetasol Propionate in Patients With Mild-moderate Plaque-type Psoriasis
Brief Title: Topical 1% Methotrexate Gel Versus Clobetasol Propionate in Patients With Psoriasis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr. Jose N. Rodriguez Memorial Hospital and Sanitarium (Other)
Responsible Party: Principal Investigator, John Benjamin B. Gochoco, Principal Investigator, Dr. Jose N. Rodriguez Memorial Hospital and Sanitarium
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: JNRodriguezMHS
Record Dates: First submitted 2024-08-07; First posted 2024-08-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Pilot Study; Psoriasis
Keywords: topical methotrexate gel; Clobetasol
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical 1% methotrexate gel (Experimental): topical 1% methotrexate gel 2x a day for 6 weeks
  Interventions: Drug: topical 1% methotrexate gel
- clobetasol propionate 0.05% ointment (Active Comparator): clobetasol propionate 0.05% ointment 2x a day for 6 weeks
  Interventions: Drug: clobetasol propionate 0.05% ointment

INTERVENTIONS:
Drug: topical 1% methotrexate gel — topical 1% methotrexate gel
  Other Names: clobetasol propionate 0.05% ointment
  Arms: topical 1% methotrexate gel
Drug: clobetasol propionate 0.05% ointment — clobetasol propionate 0.05% ointment
  Arms: clobetasol propionate 0.05% ointment

SUMMARY:
A pilot study on the formulation of topical methotrexate was conducted. Patients after baseline evaluation were randomly placed into either topical 1% methotrexate gel or clobetasol propionate 0.05% ointment which was applied for 6 weeks. PASI score was assessed at two-week intervals for a total of eight weeks. Blood chemistry parameters, whole abdomen ultrasound, and adverse drug reactions while on treatment and after eight weeks were monitored as secondary outcome measures.

DETAILED DESCRIPTION:
This is a pilot study done for a year at the dermatologic clinic of a tertiary hospital. The study was approved by the Institutional Review Board and followed the declaration of Helsinki Principles for patient rights.

Patients clinically diagnosed with psoriasis were chosen for the study. Inclusion criteria for the participants include the following: patients with stable mild-moderate plaque psoriasis, regardless of chronicity of the disease, involving less than 30% of the body surface area (BSA) with a negative pregnancy test for female participants of reproductive age. On the other hand, the exclusion criteria for the participants include the following: patients with psoriatic lesions on the face and/or scalp, administration of topical, systemic, or intralesional therapy or UV radiation therapy for at least 2 weeks before the study. Patients with deranged laboratory results at the baseline of the study, minors or lactating mothers, and patients planning a pregnancy with their spouses/partners in the next three months.

The gathered patients with psoriasis were randomly and equally divided, by a tossed coin, into two groups according to the type of treatment the participant received. Group I was treated with the MTX 1% gel while the other group was treated with clobetasol propionate 0.05% ointment. The sampling method used was complete enumeration sampling was used for patients with psoriasis from 2022 to 2023. Should the number of willing participants for the study exceed the determined sample size, only the first patients to satisfy the inclusion criteria were included in the study. The study blinded the participants, the investigators, and the statistician when it came to the treatment involved until the trial was finished.

After the patient agreed to the set guidelines of the study, photographs of the lesions, PASI score, and laboratory parameters including blood urea nitrogen (BUN), creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and whole abdomen ultrasound were taken at baseline of the study. These laboratories were once again done on week 6 at the end of the application of the assigned topical. The participants were asked to return for follow-up after two weeks of wash-out period, week 8, to see if there was sustained remission defined as no new psoriatic lesion after two weeks of discontinuation of the assigned topical medication. The procedure for this study is detailed in Figure 1.

The withdrawal criteria for the participants in the study were as follows: experienced exacerbation defined as a 125% increase of PASI from the baseline, failure to apply the medication for two consecutive days, failure to appear in one of the follow-up consultations which was done every two weeks. Appearance of adverse drug reactions such as, but not limited to: new lesions, increase in erythema, scaling, or thickening of previous lesions, and intractable pruritus. If any of the abovementioned criteria were present, the participant was asked to discontinue the use of the trial medication and was given the standard treatment therapy (topical corticosteroid) instead.

The intervention used in the study comprised of identical blue-green containers filled with either MTX 1% gel or clobetasol propionate 0.05% ointment and were given to the study participants. They were instructed to apply only to the psoriatic lesion. Participants were educated to recognize common side effects such as stings of dermatitis, irritation, and burning. Each Participant was instructed to apply the given topical formula twice daily for six weeks. No occlusion dressings were used. Avoidance to prolonged sunlight exposure as well as the use of other emollients were advised.

Primary endpoints is the BSA involved in the psoriasis lesions and PASI score. Secondary endpoints include the result of the laboratory parameters of the patient after week six and determination of noted adverse drug reactions on both treatment arms.

The PASI scores of the participants were assessed with an independent sample t-test for comparison between variables.7 Data were analyzed on Statistical Package for Social Science (SPSS) version 11. A p-value of less than 0.05 was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with stable mild-moderate plaque psoriasis, regardless of chronicity of the disease,
* involving less than 30% of the body surface area (BSA)
* negative pregnancy test for female participants of reproductive age

Exclusion Criteria:

* patients with psoriatic lesions on the face and/or scalp,
* administration of topical, systemic, or intralesional therapy or UV radiation therapy for at least 2 weeks before the study.
* Patients with deranged laboratory results at the baseline of the study, minors or lactating mothers
* patients planning a pregnancy with their spouses/partners in the next three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) score computed | 8 weeks
  Psoriasis Area and Severity Index scores range from 0 to 72. In general, the higher the PASI score, the more severe is the disease

SECONDARY OUTCOMES:
Change in baseline laboratory results | 8 weeks
  blood urea nitrogen (BUN)
Change in baseline laboratory results | 8 weeks
  creatinine
Change in baseline laboratory results | 8 weeks
  alanine aminotransferase (ALT)
Change in baseline laboratory results | 8 weeks
  aspartate aminotransferase (AST)
Change in baseline laboratory results | 8 weeks
  whole abdomen ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: John Benjamin B Gochoco, MD, Principal Investigator — Dr. Jose N. Rodriguez Memorial Hospital and Sanitarium
Locations (1):
- Dr. Jose N. Rodriguez Memorial Hospital and Sanitarium, Caloocan, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Yes
The whole study will be available
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Access to all

REFERENCES:
- [Background] Kimwell MJM, de Guzman DC, Onda AJM, Dofitas BL, Frez MLF, Mendoza CG, Rivera FD 4th, Almirol BJQ, Malaluan MJQ, Guce K. Economic Evaluation of Selected Interleukin Inhibitors Versus Methotrexate for Moderate-to-Severe Plaque Psoriasis From the Philippine Payer Perspective. Value Health Reg Issues. 2023 Mar;34:100-107. doi: 10.1016/j.vhri.2022.12.001. Epub 2023 Jan 11. PMID 36638606
- [Background] Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med. 2009 Jul 30;361(5):496-509. doi: 10.1056/NEJMra0804595. No abstract available. PMID 19641206
- [Background] Sarac G, Koca TT, Baglan T. A brief summary of clinical types of psoriasis. North Clin Istanb. 2016 Jun 14;3(1):79-82. doi: 10.14744/nci.2016.16023. eCollection 2016. PMID 28058392
- [Background] Hsu S, Papp KA, Lebwohl MG, Bagel J, Blauvelt A, Duffin KC, Crowley J, Eichenfield LF, Feldman SR, Fiorentino DF, Gelfand JM, Gottlieb AB, Jacobsen C, Kalb RE, Kavanaugh A, Korman NJ, Krueger GG, Michelon MA, Morison W, Ritchlin CT, Stein Gold L, Stone SP, Strober BE, Van Voorhees AS, Weiss SC, Wanat K, Bebo BF Jr; National Psoriasis Foundation Medical Board. Consensus guidelines for the management of plaque psoriasis. Arch Dermatol. 2012 Jan;148(1):95-102. doi: 10.1001/archdermatol.2011.1410. PMID 22250239
- [Background] Haider S, Wahid Z, Najam-Us-Saher, Riaz F. Efficacy of Methotrexate in patients with plaque type psoriasis. Pak J Med Sci. 2014 Sep;30(5):1050-3. doi: 10.12669/pjms.305.4451. PMID 25225524
- [Background] Pinto MF, Moura CC, Nunes C, Segundo MA, Costa Lima SA, Reis S. A new topical formulation for psoriasis: development of methotrexate-loaded nanostructured lipid carriers. Int J Pharm. 2014 Dec 30;477(1-2):519-26. doi: 10.1016/j.ijpharm.2014.10.067. Epub 2014 Nov 1. PMID 25445970
- [Background] Dawson, B., & Trapp, R. G. (2001). Basic et clinical biostatistics. Buch. Lange Med. Books/Mcgraw-Hill.
- [Background] Coondoo A, Phiske M, Verma S, Lahiri K. Side-effects of topical steroids: A long overdue revisit. Indian Dermatol Online J. 2014 Oct;5(4):416-25. doi: 10.4103/2229-5178.142483. PMID 25396122
- [Background] Zhou Y, Yang L, Lyu Y, Wu D, Zhu Y, Li J, Jiang D, Xin X, Yin L. Topical Delivery of ROS-Responsive Methotrexate Prodrug Nanoassemblies by a Dissolvable Microneedle Patch for Psoriasis Therapy. Int J Nanomedicine. 2023 Feb 18;18:899-915. doi: 10.2147/IJN.S394957. eCollection 2023. PMID 36824414